CLINICAL TRIAL: NCT04479709
Title: The Urinary Microbiome Before and After Treatment With Intradetrusor Onabotulinum Toxin A Injection for Overactive Bladder
Brief Title: The Urinary Microbiome in Patients Receiving Intradetrusor Botox Injections
Status: Completed | Type: Observational
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey Mangel, Associate Professor, Case Western Reserve University School of Medicine, MetroHealth Medical Center
Other Study IDs: IRB20-00120
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Overactive Bladder
Keywords: Overactive bladder; Urinary microbiome
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An altered urinary microbiome (UM) may explain the symptoms in overactive bladder (OAB) patients who were previously considered to have "idiopathic" OAB. To date, most research on the relationship between OAB and the UM has focused on differentiating between the UM of a normal bladder and that of an OAB bladder. There is currently a paucity of data on the way that OAB therapy impacts the UM. One of the few studies to evaluate the UM pre- and post-OAB treatment focused on how management with solifenacin affected the UM, but no studies have evaluated how intravesical onabotulinumtoxin A injections (IOI) affects the UM. Understanding IOI's impact on the UM is particularly interesting because despite both anticholinergics and IOI exerting antimuscarinic affects on the bladder, IOI is often successful when anticholinergics are not. This raises the question of what other mechanisms of action IOI may have in the bladders of OAB patients - one hypothesis is that it might stabilize the UM in those select patients who suffer from OAB due to an altered UM. The primary objective of this study is therefore to determine the UM profiles of OAB patients before and after treatment with IOI.

ELIGIBILITY:
Inclusion Criteria:

- Women undergoing intradetrusor botox injection with botox 100 U

Exclusion Criteria:

* Current UTI
* History of recurrent UTI
* History of antibiotic exposure for any reason (including if response is "unknown")
* Antibiotic exposure for any reason other than post-procedure prophylaxis during the four-week follow-up period.

Ages: 18 Years to 89 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women undergoing intradetrusor botox injection with botox 100 U
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Urinary Microbiome | 08/2020 - 08/2021
  To evaluate whether administration of intradetrusor botox injections for the treatment of overactive bladder results in changes to the urinary microbiome.

SECONDARY OUTCOMES:
Urinary Microbiome by response | 08/2020 - 08/2021
  To evaluate whether there are differences between responders and non-responders to intradetrusor botox injections in the pre- and post-treatment urinary microbiomes.
Urinary tract infection | 08/2020 - 08/2021
  Determine if there is a relationship between pre- or post-intradetrusor botox injection and the rate of urinary tract infection.
Adverse events | 08/2020 - 08/2021
  Adverse events from intradetrusor botox injection

CONTACTS AND LOCATIONS:
Locations (1):
- MetroHealth, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Palm KM, Abrams MK, Sears SB, Wherley SD, Alfahmy AM, Kamumbu SA, Chakraborty NN, Mahajan ST, El-Nashar SA, Henderson JW, Hijaz AK, Mangel JM, Pollard RR, Al-Shakhshir H, Retuerto MA, Steller KM, Elshaer M, Ghannoum MA, Sheyn D. The Response of the Urinary Microbiome to Botox. Int Urogynecol J. 2024 Jan;35(1):237-251. doi: 10.1007/s00192-023-05703-1. Epub 2024 Jan 2. PMID 38165444